CLINICAL TRIAL: NCT03596736
Title: Elbow Hemiarthroplasty Versus Total Elbow Arthroplasty for Irreparable Distal Humeral Fractures. A Multicenter Randomized Controlled Trial
Brief Title: Elbow Hemiarthroplasty Versus Total Elbow Arthroplasty for Irreparable Distal Humeral Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Lars Adolfsson, Prof, MD, PhD, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/342-31
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Distal Humerus Fracture
Keywords: Distal Humerus Fracture; Arthroplasty, Replacement, Elbow
MeSH Terms: conditions — Humeral Fractures, Distal | interventions — Arthroplasty, Replacement, Elbow

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Elbow Hemiarthroplasty (Experimental)
  Interventions: Procedure: Elbow Hemiarthroplasty
- Total Elbow Arthroplasty (Active Comparator)
  Interventions: Procedure: Total Elbow Arthroplasty

INTERVENTIONS:
Procedure: Elbow Hemiarthroplasty
  Arms: Elbow Hemiarthroplasty
Procedure: Total Elbow Arthroplasty
  Arms: Total Elbow Arthroplasty

SUMMARY:
Distal humeral fractures can be difficult to treat, in particular when the joint surface is affected (intra-articular fractures). If rigid internal fixation with plates and screws can be obtained it is considered to be the treatment of choice. In elderly patients, poor bone quality (osteopenia) and fragmentation of the articular surface can make rigid internal fixation non-reliable or even impossible. Total elbow arthroplasty has been shown to be of value in this type of situation. Elbow hemiarthroplasty has been proposed as an alternative to total elbow arthroplasty. The theoretical advantages as opposed to total elbow arthroplasty are: no restriction in the weight allowed to be lifted, complications related to polyethylene wear debris are avoided as there is no polyethylene liner and there is no ulna component that can loosen. Wear of the native ulna and instability are potential complications of elbow hemiarthroplasty.

The aim of this multicenter study is to test the hypothesis that elbow hemiarthroplasty gives better elbow function than total elbow arthroplasty for irreparable distal humeral fractures.

ELIGIBILITY:
Inclusion criteria

* Intra-articular distal humeral fracture with two or more displaced joint surface fragments devoid of soft tissue attachment
* Osteopenia
* Fracture deemed unsuitable for internal fixation
* Low-energy trauma
* Closed fracture
* Independent living

Exclusion criteria

* Comorbidity that affects elbow rehabilitation considerably
* Severe pre-existing elbow disease
* Concurrent injury that affects elbow rehabilitation considerably
* Pathologic fracture
* Vascular injury
* Inability to participate in follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-01-19 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire | 24 months
  The DASH questionnaire aims to assess symptoms and functional status of the upper extremities. It is a patient reported outcome measure that contains 30 core items. The score ranges from 0 to 100 points with higher scores indicating greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Adolfsson, MD, Principal Investigator — Linkoeping University
Locations (3):
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Linköping University Hospital, Linköping
  - Varberg Hospital, Varberg